CLINICAL TRIAL: NCT02887196
Title: Attitudes Toward Physical Activity and Nutrition Intervention During Cancer Treatment
Acronym: CARE
Status: Terminated | Type: Observational
Why Stopped: Saturation of a particular breast cancer treatment regimen enrolled. We will need to reexamine inclusion/exclusion criteria in future studies.
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Anne Gilmore, Assistant Professor, Pennington Biomedical Research Center
Other Study IDs: PBRC 2016-050
Record Dates: First submitted 2016-08-29; First posted 2016-09-02 (Estimated); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Breast Neoplasms; Body Weight Changes
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Body Weight Changes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and serum will be stored for future research
Oversight: Data Monitoring Committee: No

SUMMARY:
Twenty-five women will be followed through their breast cancer treatment. The women will be asked to provide their opinions and desires for lifestyle intervention at different times throughout treatment. In addition, basic clinical data will be collected . The primary goal of this pilot study is to investigate the physical and behavioral changes that occur in patients receiving treatment for breast cancer.

DETAILED DESCRIPTION:
In this cross sectional, longitudinal, observational study, 25 women will be followed through their treatment for stage I-III breast cancer. The women will be asked to provide their opinions and desires for lifestyle intervention at four timepoints throughout treatment. In addition to qualitative data, basic clinical data will be collected (anthropometrics, vital signs, dietary intake, and physical activity). The primary goal of this pilot study is to investigate the anthropometric and behavioral changes that occur in patients undergoing adjuvant chemotherapy for breast cancer.

Aim 1: To better understand patients' attitudes toward and perceived barriers to nutrition and physical activity interventions during neoplastic treatment.

Hypothesis: Patients' reported attitudes, motivation, and perceived barriers will change throughout treatment.

Aim 2: To measure the physical and metabolic changes that occur throughout neoplastic treatment for breast cancer.

Hypothesis: Over 50% of the participants will gain body weight during treatment and metabolic parameters will trend with body weight change.

ELIGIBILITY:
Inclusion Criteria:

* Female
* ≥18 years of age
* Diagnosed with stage I, II or III breast cancer with plans to undergo endocrine and/or chemotherapy treatment (radiation in combination with one or more of these therapies is acceptable)
* Willing to complete up to 4 clinic visits

Exclusion Criteria:

* Have received neoadjuvant therapy for current diagnosis
* Currently receiving adjuvant chemotherapy or other adjuvant therapy that was initiated prior to study enrollment
* History of cancer and neoplastic treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community hospitals and physician offices in the Baton Rouge, LA area
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2016-12; Primary Completion 2018-09-11 (Actual); Study Completion 2018-09-18 (Actual)

PRIMARY OUTCOMES:
Perceived attitudes towards lifestyle interventions | 9 months
  Qualitative data collected via semi-structured interview

SECONDARY OUTCOMES:
Diet | 9 months
  24 hour recall (ASA24) to assess food intake changes throughout treatment
Physical Activity | 9 months
  Wrist worn Actigraph accelerometer to assess activity changes throughout treatment
Body Weight | 9 months
  Body weight change throughout treatment

CONTACTS AND LOCATIONS:
Overall Officials: Anne Gilmore, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided